CLINICAL TRIAL: NCT00057031
Title: A Phase 2, Multicenter, Open Label Study of the Safety and Efficacy of High-Dose Pulse Administration DN-101 (Calcitriol) in Patients With Myelodysplastic Syndrome
Brief Title: Study of High-Dose Pulse Administration DN-101 (Calcitriol) in Patients With Myelodysplastic Syndrome (MDS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novacea (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: DN101-003
Record Dates: First submitted 2003-03-26; First posted 2003-04-01 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2005-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Calcitriol

INTERVENTIONS:
Drug: DN-101 (calcitriol)

SUMMARY:
The purpose of this study is to determine the safety and efficacy of DN-101 (calcitriol) in patients with myelodysplastic syndrome who are dependent on repeat blood transfusions.

DETAILED DESCRIPTION:
DN-101 is an experimental drug that has not been approved by the Food and Drug Administration (FDA). It is a newly formulated pill that contains high amounts of calcitriol, a naturally occurring hormone and the biologically active form of vitamin D. The natural vitamin D found in dairy products or in typical vitamin pills, must be chemically changed by the liver and kidney into calcitriol before it is biologically active. The body normally uses small amounts of calcitriol to regulate its blood calcium levels. However, for any possible therapeutic effect, MDS patients require much higher levels of calcitriol than the body can produce from dietary vitamin D. DN-101 provides MDS patients with high doses of calcitriol in a pill form.

Laboratory studies have demonstrated evidence supporting the use of calcitriol in MDS. High dose calcitriol slows the growth of leukemic cells (cancerous cells) and increases the growth of normal bone marrow cells. Some patients with MDS may have low levels of calcitriol in their bone marrow.

Clinical study results in patients with MDS have been mixed- some positive and some negative results. Elevated calcium in the blood occurred frequently and prevented the use of higher, more potentially therapeutic doses.

Novacea tested a new formulation of calcitriol, DN-101, in a Phase 1 study. In that study the maximum tolerated dose of DN-101 that did not cause high blood calcium levels when given weekly for several months was determined. That dose is within the range that is potentially therapeutic for MDS patients and will be used in this MDS study.

The purposes of this study are to determine if HDPA DN-101 treatment:

* increases the number of red blood cells, white blood cells, and platelets in the blood
* reduces the number of blood transfusions
* reduces the number of serious infections requiring antibiotics
* reduces the number of serious bleeding events
* improves fatigue

ELIGIBILITY:
* Diagnosis of low or intermediate-1 risk MDS
* Dependent on monthly blood transfusions
* No cancer within the last 5 years (cured skin cancer is allowed)
* No heart attack or stroke within the last 6 months
* No kidney stones within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2002-11; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - University of California, San Francisco, San Francisco, California
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Rush Cancer Institute MDS Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Cleveland Clinic Foundation, Taussig Cancer Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Boston Baskin Cancer Group, Memphis, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Mellibovsky L, Diez A, Perez-Vila E, Serrano S, Nacher M, Aubia J, Supervia A, Recker RR. Vitamin D treatment in myelodysplastic syndromes. Br J Haematol. 1998 Mar;100(3):516-20. doi: 10.1046/j.1365-2141.1998.00598.x. PMID 9504634
- [Background] Beer TM, Munar M, Henner WD. A Phase I trial of pulse calcitriol in patients with refractory malignancies: pulse dosing permits substantial dose escalation. Cancer. 2001 Jun 15;91(12):2431-9. PMID 11413535
- [Background] Beer TM, Eilers KM, Garzotto M, Egorin MJ, Lowe BA, Henner WD. Weekly high-dose calcitriol and docetaxel in metastatic androgen-independent prostate cancer. J Clin Oncol. 2003 Jan 1;21(1):123-8. doi: 10.1200/jco.2003.05.117. PMID 12506180